CLINICAL TRIAL: NCT05923918
Title: A Prospective, Randomized, Parallel, Multi-center, Phase 3 Trial to Evaluate Safety and Efficacy of PBK_M2101
Brief Title: A Study to Evaluate Safety and Efficacy of PBK_M2101
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PBK_M2101_301
Record Dates: First submitted 2023-05-18; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Intestinal Disease; Colonic Diseases; Gastrointestinal Disease; Digestive System Disease
MeSH Terms: conditions — Intestinal Diseases; Colonic Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — Sulfates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- test 1 (Experimental): PBK_M2101, 2-Day Regimen
  Interventions: Drug: PBK_M2101 2-Day
- test 2 (Experimental): PBK_M2101, 1-Day Regimen
  Interventions: Drug: PBK_M2101 1-Day
- active Comparator (Active Comparator): active Comparator, 2-Day Regimen
  Interventions: Drug: Oral Sulfate Tablet 2-Day

INTERVENTIONS:
Drug: PBK_M2101 2-Day — Subjects who are randomized into group test 1 will receive bowel preparation from evening to next morning.
  Arms: test 1
Drug: PBK_M2101 1-Day — Subjects who are randomized into group test 2 will receive bowel preparation on the same-day.
  Arms: test 2
Drug: Oral Sulfate Tablet 2-Day — Subjects who are randomized into group active comparative will receive bowel preparation from evening to next morning.
  Arms: active Comparator

SUMMARY:
This clinical trial was prospective, randomized, single-blind, 3-treatment arm, parallel treatment group, and active-controlled. , Multi-center, Phase 3 confirmatory clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is informed and give a consent in voluntary
* Patients who is scheduled a esophagogastroduodenoscopy and colonoscopy
* BMI 19≤and<30

Exclusion Criteria:

* Patients who participate in other interventional study or had participated within 30 days before screening
* Pregnant or breast-feeding women who do not want to stop breast-feeding
* Uncontrolled hypertension
* Uncontrolled diabetes
* Fluid or electrolyte (Na, K, Ca, Mg, chloride, bicarbonate) disturbance
* HIV infection and/or chronic hepatitis B or C
* Patients who has a difficulty to participate because of severe nausea or vomiting
* History of colon surgery and abdominal surgery within 6 month; need an emergency surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Successful cleansing rate | From day of first dosing to day of colonoscopy
  %Patient with HCS-graded A or B

SECONDARY OUTCOMES:
Overall cleansing rate | From day of first dosing to day of colonoscopy
  %Patient with each HCS-grade (A, B, C, D)
Mean segmental cleansing score | From day of first dosing to day of colonoscopy
  5 Segment: Rectum, Sigmoid colon, Descending colon, Transverse colon, Ascending colon/cecum.
Mean cecal intubation time | From day of first dosing to day of colonoscopy
Mean colonoscopy withdrawal time | From day of first dosing to day of colonoscopy
Treatment compliance | From day of first dosing to day of colonoscopy
  Dosage taken/Dosage scheduled
Patient satisfaction | From day of first dosing to day of colonoscopy
  Subject questionnaire (Taste, Difficulty, Ease of taking)
Polyp detection rate | From day of first dosing to day of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Byeon, M.D., Principal Investigator — Seoul Asan Medical Center
Locations (1):
- Seoul Asan Medical Center, Seoul, South Korea